CLINICAL TRIAL: NCT05122026
Title: Safety and Tolerability of 1 Month Daily (1HP) and 3 Months Weekly (3HP) Isoniazid and Rifapentine With Pharmacokinetics of Dolutegravir (DTG) in Pregnant People With HIV
Acronym: DOLPHIN Moms
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Johns Hopkins University (Other); Weill Medical College of Cornell University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00299011; 3HP-MOMS-AUR1-6-351 (Other: The Aurum Institute)
Record Dates: First submitted 2021-10-26; First posted 2021-11-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HIV Seropositivity; Pregnancy; Tuberculosis Infection
Keywords: Dolutegravir; 3HP; Rifapentine; pharmacokinetic; TB preventive treatment
MeSH Terms: conditions — HIV Seropositivity; Latent Tuberculosis | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive either 1HP or 3HP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: One month of daily isoniazid and rifapentine (4 weeks) (Experimental): * DTG 50 mg orally BID
    * DTG 50 mg + 2 NRTI each morning (non-study)
    * 2nd dose: DTG 50 mg each evening (during 1HP)
  * 1HP: INH 300 mg + RPT 600 mg each morning for 4 weeks
  Interventions: Drug: Rifapentine; Drug: Isoniazid
- Arm 2: Three months of once-weekly isoniazid and rifapentine (12 weeks) (Experimental): * DTG 50 mg orally BID
    * DTG 50 mg + 2 NRTI each morning (non-study)
    * 2nd dose: DTG 50 mg each evening (during 3HP)
  * 3HP: INH 900 mg + RPT 900 mg each week for 12 weeks
  Interventions: Drug: Rifapentine; Drug: Isoniazid

INTERVENTIONS:
Drug: Rifapentine — As included in arm/group description
  Other Names: Priftin
Drug: Isoniazid — As included in arm/group description
  Other Names: Winthrop Isoniazid

SUMMARY:
Open-label, two-arm, randomized multicenter study to investigate the safety, tolerability, and pharmacokinetics (PK), and potential interactions between dolutegravir (DTG) and rifapentine (RPT) during pregnancy in people with HIV when RPT is given with isoniazid (INH) daily for 4 weeks (1HP) or weekly for 3 months (3HP) as part of tuberculosis (TB) preventive therapy (TPT). Adults (age ≥18) who are pregnant with a singleton pregnancy (confirmed by ultrasound) at a gestational age of 20-34 weeks and virally suppressed on an existing DTG-based plus two nucleoside reverse transcriptase inhibitors (NRTI) antiretroviral (ART) regimen for at least four weeks may participate.

DETAILED DESCRIPTION:
Enrolled participants will be randomized 1:1 to Arms 1 and 2.

Arm 1: 1HP (n=126):

Participants will start twice-daily DTG on Day 0, and will receive once-daily HP for 28 total doses, starting on Day 1. HIV viral load (VL) will be measured at baseline (screening), week 3 (Day 17), at delivery, and post-partum week 12. Safety labs: complete blood count (CBC), urea and electrolytes (U&E), creatinine, prothrombin time and international normalized ratio (PT/INR), and liver function tests (LFT) will be obtained at screening for everyone and at follow-up visits, if clinically indicated; CBCs and LFTs will be checked at delivery in all participants.

The first 25 participants enrolled to Arm 1 who consent to be in a PK substudy will participate in sparse PK blood collections for DTG. Sparse PK sampling for DTG will be performed on the morning of Day 1, before starting 1HP and before the morning dose of DTG. Additional sparse PK sampling for DTG will be performed prior to DTG dosing on Day 17 (to track with 72 hours after the 3rd dose of HP in Arm 2).

A plasma specimen for RPT PK will also be collected on Day 17.

Arm 2: 3HP (n=126):

Participants will start twice-daily DTG on Day 0, and will receive once-weekly HP for 12 total doses starting on Day 1. HIV VL will be measured at baseline (screening), week 3 (Day 17), at delivery, and at post-partum week 12. Safety labs: CBC, U&E, creatinine, PT/INR, and LFTs will be obtained at screening for everyone and at follow-up visits, if clinically indicated; CBCs and LFTs will be drawn at delivery.

The first 25 participants enrolled to Arm 2 who consent to be in a PK substudy will participate in sparse PK blood collections for DTG. Sparse PK sampling for DTG will be performed on the morning of Day 1, before starting 3HP, and before the morning dose of DTG. Additional sparse PK sampling for DTG will be performed on Day 17 prior to DTG dosing (72 hours after the 3rd dose of HP) and on Day 52 prior to DTG dosing (72 hours after the 8th dose of HP).

There will not be plasma collection on Day 17 for RPT PK in Arm 2, because specimen collection would be 72 hours after the weekly HP dose and a RPT level will likely not be detectable.

Interim analysis will occur when 25 participants each from Arms 1 and 2 have completed the Week 3 (Day 17) sparse PK visit. Ongoing enrolment will not be paused during the interim analysis, which will assess DTG PK, safety, and VL data.

Enrollment will be paused if accrual to each arm reaches 101 participants before the interim analysis has been completed. Once results are available, then enrollment will restart with dosing (daily vs. BID) based on the DTG PK results.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Weight > 50 kg
3. Documented HIV infection
4. At least 4 weeks of ART and virally suppressed on dolutegravir plus two NRTIs
5. Undetectable HIV-1 viral load
6. Pregnancy at 20-34 weeks as confirmed by ultrasound
7. Singleton pregnancy

Exclusion Criteria:

1. Confirmed or suspected TB disease
2. Likely to move from the study area during the study period
3. Known exposure to pulmonary TB cases with known or suspected resistance to isoniazid or rifampicin in the source case
4. TB treatment within the past year
5. TB preventive therapy within the last year
6. Sensitivity or intolerance to isoniazid or rifamycins
7. On nevirapine, etravirine, rilpivirine, PI-based, or raltegravir-containing ART regimens
8. Suspected acute hepatitis or known chronic liver disease; HBsAg positivity; severe hepatic impairment
9. Alanine aminotransferase (ALT) ≥ 3 times the upper limit of normal (ULN)
10. Total bilirubin ≥ 2.5 times the ULN
11. Absolute neutrophil count (ANC) < 750 cells/mm3
12. Creatinine clearance < 50 ml/min
13. Self-reported alcohol use exceeding 21 units per week
14. Karnofsky status < 80
15. On prohibited medications e.g. dofetilide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | from study entry at Week 0 through post partum Week 24, to be reported at end of trial
  Maternal all-cause mortality (both groups)
Targeted serious adverse events (SAEs) | from study entry at Week 0 through post partum Week 12, to be reported at end of trial
  Premature discontinuation for toxicity or intolerance, Grade 3 or higher maternal bleeding, peripheral neuropathy, elevated LFTs), targeted pregnancy outcomes (fetal demise, stillbirth, preterm delivery (PTD) <32 weeks, birthweight (BW) <1500g, neonatal death <28 days of age), or permanent discontinuation due to toxicity (both groups)
PK sampling of Dolutegravir - Cl/F parameter | PK sampling at Week 1 (Day 1) and Week 3 (Day 17) for both groups, and at Week 8 (Day 52) for Group 2 (3HP arm), to be reported at end of trial
  Oral clearance in the presence or absence of 1HP or 3HP (both groups)
PK sampling of Dolutegravir - AUC parameter | PK sampling at Week 1 (Day 1) and Week 3 (Day 17) for both groups, and at Week 8 (Day 52) for Group 2 (3HP arm), to be reported at end of trial
  Area under the plasma drug concentration-time curve (AUC) in the presence or absence of 1HP or 3HP (both groups)
PK sampling of Dolutegravir - Ctau parameter | PK sampling at Week 1 (Day 1) and Week 3 (Day 17) for both groups, and at Week 8 (Day 52) for Group 2 (3HP arm), to be reported at end of trial
  Trough concentration (Ctau) in the presence or absence of 1HP or 3HP (both groups)

SECONDARY OUTCOMES:
HIV-1 RNA viral load- maternal | HIV viral load to be measured at Screening, Week 3, at Delivery, and post partum Week 12, to be reported at end of trial
  Maternal HIV-1 RNA viral load (copies/ml) (both groups)
DTG Dose selection | Dose selection will be determined at the interim analysis to be conducted when 25 participants from Arms 1 and 2 respectively have completed the Week 3 PK visit. Based upon these results, new enrollees will receive DTG either once or twice daily.
  Dose options for DTG with 1HP or 3HP derived by simulation using nonlinear mixed effects models (both groups)
PK sampling of RPT - AUC parameter | PK sampling at Week 3 (Day 17 ) to be reported at end of trial
  Area under curve (AUC) in participants taking 1HP (Group 1)
PK sampling of RPT - Ctau parameter | PK sampling at Week 3 (Day 17 ) to be reported at end of trial
  Trough concentration (Ctau) in participants taking 1HP (Group 1)
Adverse Events- maternal | from study entry at Week 0 through post partum Week 12, to be reported at end of trial
  Grade 3 or higher maternal adverse events (AE) (all groups)
Adverse Events- pregnancy | from study entry at Week 0 through post partum Week 12, to be reported at end of trial
  Grade 3 or higher pregnancy adverse events (AE) (all groups)
Adverse Events- infant | from Delivery through post partum Week 24, to be reported at end of trial
  Grade 3 or higher infant adverse events (AE) (all groups)
HIV infection- infant | from Delivery through post partum Week 24, to be reported at end of trial
  Infant HIV infection (all groups)
Infant growth parameters- HAZ | from Delivery through post partum Week 24, to be reported at end of trial
  Height-for-age z-score (all groups)
Infant growth parameters- WAZ | from Delivery through post partum Week 24, to be reported at end of trial
  Weight-for-age z-score (WAZ) (all groups)
Infant growth parameters- HCAZ | from Delivery through post partum Week 24, to be reported at end of trial
  Head circumference-for-age z-score (HCAZ) (all groups)
TB disease-maternal | from study entry at Week 0 through post partum Week 24, to be reported at end of trial
  confirmed maternal TB disease (all groups)
TB disease-infant | from Delivery through post partum Week 24, to be reported at end of trial
  confirmed or suspected infant TB disease (all groups)
Treatment adherence- HP | from study entry at Week 0 through up to 8 weeks of 1HP (Group 1) or up to 16 weeks of 3HP (Group 2) , to be reported at end of trial
  Proportion of doses taken for 1HP and 3HP regimens

CONTACTS AND LOCATIONS:
Overall Officials: Dr Vaneshree Govender, Principal Investigator — Aurum Institute
Locations (3):
- South Africa (3):
  - FAMily Centre for Research with Ubuntu (FAMCRU), Cape Town, Cape Town
  - The Aurum Institute: Tembisa Clinical Research Centre, Tembisa, Gauteng
  - Peri Natal HIV Research Unit - Klerksdorp Tshepong Hospital, Klerksdorp, North West

IPD SHARING:
Plan to Share IPD: No